CLINICAL TRIAL: NCT04652830
Title: Randomised Controlled Trial to Assess the Benefit of Naprapathy Training for Preventing Problems from Rectus Abdominis Diastasis
Brief Title: Naprapathy Training for Postpartum DRAM Prevention
Acronym: NapraDRAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Hela Kvinnans Klinik (Unknown)
Responsible Party: Principal Investigator, Gabriel Sandblom, Research group leader, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NapraDRAM
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Diastasis Recti
Keywords: Diastasis Recti; Naprapathy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Single-blinded parallel randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors performing the follow-up ultrasound and clinical examination are blinded to the allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naprapathy training (Active Comparator): Training program for three months
  Interventions: Behavioral: Naprapathy training
- Control group (Placebo Comparator): No change of daily routines
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Naprapathy training — Active training aimed at strengthening the abdominal muscles
  Arms: Naprapathy training
Other: Control group — No change of daily routines in regard to training
  Arms: Control group

SUMMARY:
A randomised controlled trial with the aim of analysing the effectiveness of a training program intended to prevent symptoms related to DRAM in the postpartum period.

DETAILED DESCRIPTION:
Diastasis of the rectus abdominis muscles (DRAM) is a common condition after pregnancy and after great loss of weight. Distension of linea alba is a normal process during pregnancy caused by the growing fetus as well as from hormonal changes.

In the majority of cases, DRAM regresses during the postpartum period and the abdomen resumes its normal function. I some cases, however, the DRAM persists for a long period. This may result in trunk instability, back pain and decreased abdominal muscle strength. Risk factors for persisting DRAM are multiparity, high maternal age and cesarean delivery.

Little is known about how DRAM affects abdominal function. The lack of studies on the impact of DRAM on trunk instability and back pain has made it difficult to evaluate studies aiming at reducing the problems caused by DRAM.

Conservative management, including training aiming at strengthening the abdominal muscles, is usually considered the first hand alternative. There are, however, few studies on the effectiveness of training programs for the purpose of preventing DRAM.

The purpose of the present trial is to evaluate the effectiveness of a specific training program during a limited period of time postpartum in women with DRAM. The investigators also intend to study the changes in anatomy of linea alba during the postpartum period and explore whether the changes are affected by the training.

The study will be conducted as a randomized single-blind controlled trial. Women with diastasis of > 3 cm will be invited. The aim is to include 70 women. Half of them will be randomized to a training program for 3 month and the other half will be followed as a control group.

At the start of the study, the line alba is examined with ultrasound. The width of the diastasis is registered. The laxity and thickness of line alba are also evaluated. The abdominal circumference is measured at rest and under straining, in different postures.

At the start of the study, the woman is request to rate her level of physical activity (Baecke questionnaire) pain, self-assessed functional level (DRI), back pain (Oswestry low back disability index), urinary incontinence (UDI-6, IID-7) and quality of life (EQ-5D). The Abdominal Trunk Function Protocol (ATFP) is also registered at the start.

The assessors performing the ultrasound examination and physical examinations are blinded to the allocation. Women allocated to the training program perform exercises with a duration of ten minutes 6 days a week. They also perform 3 exercises with a duration of 60 seconds three times a day. The exercises are continued for three months. All women, those allocated to training as well as the control group, are invited to follow-up examinations 6 and 12 months after inclusion.

At both follow-up examinations the abdominal wall is investigated with ultrasound, the abdominal circumference is measured and the woman is requested to respond to all the questionnaires that she received at the start of the study.

Analyses will focus on the effect of the training program on the width and laxity of the linea alba as well as symptoms of back pain, trunk instability and incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Uni- and multiparous women 3-12 months postpartum
* Ability to understand Swedish language
* Ability participate in a three months follow-up program
* Diastasis of the rectus abdominis muscles > 3 cm

Exclusion Criteria:

* Ongoing pregnancy
* Age <18 years or >50 years
* < 3 months or >12 months post partum
* History of neurologic, musculoskeletal or psychiatric disorders
* Interrectal diastasis < 3 cm

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only females after childbirth
Enrollment: 70 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Abdominal Trunk Function | One year
  Abdominal Trunk Function assessed with the Abdominal Trunk Function Protocol (ATFP). Six separate subscales.

SECONDARY OUTCOMES:
Disability | One year
  Disability rated with the Disability Rating index (DRI). Rates ranging from 0 to 1200, where high ratings indicate worse outcome.
Urinary Incontinence | One year
  Urinary incontinence rated with UDI-6 (urinary distress inventory). Rates ranging from 0 to 18, where high rates indicate worse outcome.
Health-related Quality of Life | One year
  Quality of Life rated with EQ-5D
Width of the diastasis | One year
  Width measured with ultrasound
Linea alba distortion index | One year
  Distortion of the linea alba at rest and under tension assessed with ultrasound. Distortion index: average deviation of the LA from the shortest path between the recti, ranging from 0 to 1, higher index indicating greater distortion.
Urinary incontinence | One year
  Incontinence symptoms rated with the IID-7 (incontinence impact questionnaire). Rates ranging from 0 to 21, where high rates indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Sandblom, Ass Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Hela Kvinnans Klinik, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No